CLINICAL TRIAL: NCT01586286
Title: Does Adjunctive Treatment With Vaginal Nifedipine Result in Symptomatic Improvement in Patients With Levator Myalgia and Pelvic Floor Pain Who Are Undergoing Pelvic Floor Physical Therapy?
Brief Title: A Study Examining the Use of Vaginal Nifedipine With Pelvic Floor Physical Therapy for Levator Myalgia and Pelvic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients were recruited over a 12 month period
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Daniel Biller, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 111573
Record Dates: First submitted 2012-04-20; First posted 2012-04-26 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Levator Ani Syndrome
Keywords: Levator Myalgia; Pelvic Pain; Vaginismus; Myofascial pain syndromes
MeSH Terms: conditions — Levator syndrome; Pelvic Pain; Vaginismus; Myofascial Pain Syndromes | interventions — Nifedipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ointment Base (Placebo Comparator): Patients in this arm will serve as the control and will undergo pelvic floor physical therapy and receive placebo (lanolin and mineral oil base).
  Interventions: Drug: Placebo Ointment Base
- Nifedipine Ointment (Active Comparator): Patients in this arm will undergo pelvic floor physical therapy, but will receive compounded vaginal nifedipine.
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine — Nifedipine - 0.2% concentration in a lanolin base; administered twice per day for 28 days; as a vaginal ointment applied to vulvar and vaginal area
  Arms: Nifedipine Ointment
Drug: Placebo Ointment Base — Placebo administered twice per day for 28 days; as a vaginal ointment applied to vulvar and vaginal area
  Arms: Ointment Base

SUMMARY:
The objective of this study is to perform a randomized controlled trial among female patients with a diagnosis of pelvic floor hypertonus (extreme muscle tension) with associated pain, dysfunctional voiding, dyspareunia, and/ or obstructed defecation.

DETAILED DESCRIPTION:
Given the paucity of information and the magnitude of debilitation that can be associated with chronic pain syndromes, the potential to ameliorate pain and successfully treat these symptoms is an area that merits further exploration. In this study, we hypothesize that the addition of vaginal nifedipine to a physical therapy protocol will result in greater treatment success than treatment with physical therapy alone.

The objective is to perform a randomized controlled trial among female participants with a diagnosis of pelvic floor hypertonus with associated pain, dysfunctional voiding, dyspareunia, and/or obstructed defecation. Group 1 will serve as the control and will undergo pelvic floor physical therapy and placebo (lanolin and mineral oil base). Group 2 will also undergo pelvic floor physical therapy, but will receive compounded vaginal nifedipine.

Specific aims include:

1. Comparison of subjective outcome measures, specifically quality of life metrics scales: Pelvic Floor Distress Inventory, Pelvic Floor Impact Questionnaire, and validated 11-point pain scale.
2. Comparison of objective outcome measures, specifically a validated digital assessment of pelvic floor strength: the Oxford scale.

Group 1 will serve as the control and will undergo pelvic floor physical therapy and placebo (lanolin base). Group 2 will also undergo pelvic floor physical therapy, but will receive compounded vaginal nifedipine. We will collect data on these patients to determine if the treatment of vaginal nifedipine with physical therapy provides a more successful treatment for this pelvic floor dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Subject has levator myalgia upon appropriate pelvic exam that reproduces HPI pain
* Subject has symptoms such as voiding dysfunction, dyspareunia, vaginismus, or obstructed defecation
* Subject is willing and able to give written consent for the study
* Subject is willing to undergo treatment with pelvic physical therapy & vaginal nifedipine
* Subject is able to speak, read, and write in English
* Subject is at least 18 years of age

Exclusion Criteria:

* Subject has previously diagnosed interstitial cystitis
* Subject has an active case of symptomatic HSV, syphilis, or shingles
* Subject has a history of uncontrolled hypertension
* Subject is already taking a calcium channel blocker
* Subject has a history of MI, CHF, or arrhythmia
* Subject has a history of neurologic disease
* Subject has a history of congenital or progressive musculoskeletal disease
* Subject has a history of bladder or pelvic cancer and/or pelvic radiation
* Subject is planning to be or currently pregnant
* Subject has known allergy or adverse reaction to nifedipine
* Subject has known allergy or adverse reaction to lanolin, mineral oil, petrolatum
* Subject is undergoing pharmacologic treatment specific to pelvic pain
* Subject is taking oral beta adrenergic antagonist medication
* Subject has an active pelvic or vaginal infection
* Subjects with hypotension on screening physical examination (i.e. confirmed SBP<90 mmHg or DBP<60 mmHg).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Improvement in Quality of Life | To be assessed 1 month post-treatment.
  The primary outcome will measure quality of life metrics, as reported by the patient herself. We will use the following validated instruments: Pelvic Floor Distress Inventory, Pelvic Floor Impact Questionnaire, and validated 11-point pain scale. The aim is to measure whether the patient experienced improvement in her symptoms when vaginal nifedipine was administered (in addition to physical therapy).

SECONDARY OUTCOMES:
Improvement in Hypertonic Pelvic Floor Muscles | To be assessed at baseline and the following post-treatment intervals: 1, 2, 3, and 6 months
  The secondary outcome measure will be assessed and reported by the healthcare provider at the above visits. After instructing the patient to voluntarily relax the pelvic floor muscles, the resting tone will be measured using the Oxford scale, which is a validated digital assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Biller, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Mathias SD, Kuppermann M, Liberman RF, Lipschutz RC, Steege JF. Chronic pelvic pain: prevalence, health-related quality of life, and economic correlates. Obstet Gynecol. 1996 Mar;87(3):321-7. doi: 10.1016/0029-7844(95)00458-0. PMID 8598948
- [Background] Reiter RC. A profile of women with chronic pelvic pain. Clin Obstet Gynecol. 1990 Mar;33(1):130-6. No abstract available. PMID 2178830
- [Background] Butrick CW. Pelvic floor hypertonic disorders: identification and management. Obstet Gynecol Clin North Am. 2009 Sep;36(3):707-22. doi: 10.1016/j.ogc.2009.08.011. PMID 19932423
- [Background] Rosenbaum TY, Owens A. The role of pelvic floor physical therapy in the treatment of pelvic and genital pain-related sexual dysfunction (CME). J Sex Med. 2008 Mar;5(3):513-23; quiz 524-5. doi: 10.1111/j.1743-6109.2007.00761.x. PMID 18304280
- [Background] Onghena P, Van Houdenhove B. Antidepressant-induced analgesia in chronic non-malignant pain: a meta-analysis of 39 placebo-controlled studies. Pain. 1992 May;49(2):205-219. doi: 10.1016/0304-3959(92)90144-Z. PMID 1535121
- [Background] Bornstein J, Tuma R, Farajun Y, Azran A, Zarfati D. Topical nifedipine for the treatment of localized provoked vulvodynia: a placebo-controlled study. J Pain. 2010 Dec;11(12):1403-9. doi: 10.1016/j.jpain.2010.03.016. Epub 2010 May 26. PMID 20537958
- [Background] Katsinelos P, Papaziogas B, Koutelidakis I, Paroutoglou G, Dimiropoulos S, Souparis A, Atmatzidis K. Topical 0.5% nifedipine vs. lateral internal sphincterotomy for the treatment of chronic anal fissure: long-term follow-up. Int J Colorectal Dis. 2006 Mar;21(2):179-83. doi: 10.1007/s00384-005-0766-x. Epub 2005 Aug 10. PMID 16091912
- [Background] Nelson R. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2006 Oct 18;(4):CD003431. doi: 10.1002/14651858.CD003431.pub2. PMID 17054170
- [Background] Hundley AF, Wu JM, Visco AG. A comparison of perineometer to brink score for assessment of pelvic floor muscle strength. Am J Obstet Gynecol. 2005 May;192(5):1583-91. doi: 10.1016/j.ajog.2004.11.015. PMID 15902162